CLINICAL TRIAL: NCT04645212
Title: A Long-term Study of ADVM-022 in Neovascular (Wet) AMD - OPTIC Extension
Brief Title: Long-term Study of ADVM-022 in Neovascular (Wet) AMD [OPTIC-EXT]
Status: Active, not recruiting | Type: Observational
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADVM-022-07
Record Dates: First submitted 2020-11-20; First posted 2020-11-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Wet Age-related Macular Degeneration; Neovascular Age-related Macular Degeneration
Keywords: Choroidal Neovascularization; ADVM-022; OPTIC Study; CNV; ADVM-022-01; ADVM-022-07; AAV.7m8; Anti-VEGF therapy; Blindness; Gene therapy; Aflibercept (Eylea); Age-Related Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases; AAV Vector; Adverum; wAMD; AMD; wet AMD; nAMD; OPTIC Extension; OPTIC-EXT; Long-term Follow Up; Long-term Extension; AAV; Ixoberogene soroparvovec; Ixo-vec; Neovascular age-related macular degeneration; Adeno-associated viruses; Eye disease
MeSH Terms: conditions — Choroidal Neovascularization; Blindness; Macular Degeneration; Wet Macular Degeneration; Retinal Degeneration; Retinal Diseases; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants with wet AMD who received any dose of ADVM-022 in a prior clinical study.
  Interventions: Biological: ADVM-022

INTERVENTIONS:
Biological: ADVM-022 — Long term follow-up of subjects that received ADVM-022
  Other Names: AAV.7m8-aflibercept

SUMMARY:
ADVM-022-07 is an observational long-term extension (OPTIC-EXT) study assessing safety and efficacy of ADVM-022 gene therapy product, in participants with neovascular, or exudative (wet), age-related macular degeneration (nAMD).

DETAILED DESCRIPTION:
ADVM-022 (AAV.7m8-aflibercept) is a gene therapy product developed for the treatment of neovascular (wet) age-related macular degeneration (wet AMD). Wet AMD is a serious condition and the leading cause of blindness in the elderly. The available therapies for treating wet AMD require life-long intravitreal (IVT) injections every 4-12 weeks to maintain efficacy. A one-time IVT administration of ADVM-022 has the potential to treat wet AMD by providing durable expression of therapeutic levels of intraocular anti-VEGF protein (aflibercept) and maintaining the vision of patients. ADVM-022 is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with wet AMD receiving anti-VEGF therapy in clinical practice.

ADVM-022-07 is an observational long-term extension (OPTIC-EXT) study assessing safety and efficacy of ADVM-022 gene therapy product in participants with neovascular or exudative (wet), age-related macular degeneration (nAMD) previously treated in the OPTIC parent study (Clinical Protocol No. ADVM-022-01 [OPTIC] - NCT03748784). There is no investigational treatment administered in this study.

In Part 1 of the OPTIC-EXT study participants will roll over from the OPTIC parent study and will be followed for 3 additional years (following 2-years of assessment period in the OPTIC parent study). In Part 2 of the OPTIC-EXT study consenting participants will have 5 annual in-clinic assessments for an additional 5 years of long-term follow-up following the completion of OPTIC-EXT (Part 1). As such participants who complete the parent study as well as Part 1 and Part 2 of the OPTIC-EXT study will have had 10 years of total long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received a single dose of ADVM-022 at any dose in the OPTIC study
* Willing and able to provide informed consent

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Participants who received ADVM-022 at any dose in the OPTIC study
  * Up to 30 participants from all cohorts of OPTIC
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2030-06-26 (Estimated); Study Completion 2030-06-26 (Estimated)

PRIMARY OUTCOMES:
Severity and incidence of ocular and systemic adverse events (AEs). | 416 weeks (8 years)
  Severity and incidence of ocular and systemic adverse events

SECONDARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) from baseline, over time | 416 weeks (8 years)
  Mean change in best corrected visual acuity (BCVA) from baseline, over time
Mean change in central subfield thickness (CST) and macular volume from baseline, over time | 416 weeks (8 years)
  Mean change in central subfield thickness (CST) and macular volume from baseline, over time
Mean number of supplemental aflibercept injections over time | 416 weeks (8 years)
  Mean number of supplemental aflibercept injections over time
Percentage of participants requiring supplemental bolus aflibercept over time | 416 weeks (8 years)
  Percentage of participants requiring supplemental bolus aflibercept over time
Time to first supplemental aflibercept requirement | 416 weeks (8 years)
  Time to first supplemental aflibercept requirement
Percentage of participants without intraretinal fluid (IRF) by spectral domain optical coherence tomography (SD-OCT), over time | 416 weeks (8 years)
  Percentage of participants without intraretinal fluid (IRF) by spectral domain optical coherence tomography (SD-OCT), over time
Percentage of participants without subretinal fluid (SRF) by SD-OCT over time | 416 weeks (8 years)
  Percentage of participants without subretinal fluid (SRF) by SD-OCT over time
Time to first dry retina (defined as no IRF or SRF by SD-OCT) | 416 weeks (8 years)
  Time to first dry retina (defined as no IRF or SRF by SD-OCT)
Duration of fluid free status (defined as no IRF or SRF by SD-OCT) | 416 weeks (8 years)
  Duration of fluid free status (defined as no IRF or SRF by SD-OCT)
Percentage of participants developing geographic atrophy over time (as assessed by multiple imaging modalities) | 416 weeks (8 years)
  Percentage of participants developing geographic atrophy over time (as assessed by multiple imaging modalities)
Growth of geographic atrophy over time, as assessed by multiple imaging modalities | 416 weeks (8 years)
  Growth of geographic atrophy over time, as assessed by multiple imaging modalities
Percentage of participants with CST fluctuations > 50 μm over time | 416 weeks (8 years)
  Percentage of participants with CST fluctuations > 50 μm over time

CONTACTS AND LOCATIONS:
Overall Officials: OPTIC-EXT Medical Monitor, Study Director — Adverum Biotechnologies, Inc.
Locations (9):
- United States (9):
  - Adverum Clinical Site, Bakersfield, California
  - Adverum Clinical Site, Beverly Hills, California
  - Adverum Clinical Site, Lakewood, Colorado
  - Adverum Clinical Site, Deerfield Beach, Florida
  - Adverum Clinical Site, Reno, Nevada
  - Adverum Clinical Site, Philadelphia, Pennsylvania
  - Adverum Clinical Site, Nashville, Tennessee
  - Adverum Clinical Site, Bellaire, Texas
  - Adverum Clinical Site, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No